CLINICAL TRIAL: NCT01786057
Title: The Effect of Extracorporeal Shock Wave Therapy (ESWT)of Gastrosoleus Trigger Points in Patients With Plantar Fasciitis
Brief Title: Effect of Extracorporeal Shock Wave Therapy of Gastrosoleus Trigger Points in Patients With Plantar Fasciitis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farnaz Dehgan Hosseinabadi, Dr., Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13914022
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extracorporeal shock wave therapy 1 (Active Comparator): Extracorporeal shock wave therapy , (3000 shock waves/session of 0.2 mJ/mm2) for heel region and (400 shock waves/session of 0.2 mJ/mm2 per each trigger point) for gastrosoleus trigger points , 3 sessions at weekly intervals
  Interventions: Procedure: Extracorporeal shock wave therapy 1
- Extracorporeal shock wave therapy 2 (Placebo Comparator): Extracorporeal shock wave therapy , (3000 shock waves/session of 0.2 mJ/mm2) for heel region , 3 sessions at weekly intervals
  Interventions: Procedure: Extracorporeal shock wave therapy 2

INTERVENTIONS:
Procedure: Extracorporeal shock wave therapy 1 — Extracorporeal shock wave therapy , (3000 shock waves/session of 0.2 mJ/mm2) for heel region and (400 shock waves/session of 0.2 mJ/mm2 per each trigger point) for gastrosoleus trigger points , 3 sessions at weekly intervals
  Arms: Extracorporeal shock wave therapy 1
Procedure: Extracorporeal shock wave therapy 2 — Extracorporeal shock wave therapy , (3000 shock waves/session of 0.2 mJ/mm2) for heel region , 3 sessions at weekly intervals
  Arms: Extracorporeal shock wave therapy 2

SUMMARY:
Plantar fasciitis is one of the most common causes of heel pain. This study will be performed in the purpose of determination the effects of extracorporeal shock wave therapy of gastrosoleus trigger points in patients with plantar fasciitis

DETAILED DESCRIPTION:
Plantar fasciitis is the most common cause of inferior heel pain, A great variety of therapies have been reported for the treatment of plantar fasciitis including extracorporeal shock wave therapy. Gastrosoleus muscle dysfunction is one of the most common contributing factors to this disease .Despite the long history and the fact that this is a common diagnosis made in clinical practice, the exact cause and best treatment for this condition still are being explored. Although there is lack of high-quality studies demonstrating the efficacy of extracorporeal shock wave therapy of gastrosoleus trigger points in patients with plantar fasciitis , this study will be performed to examine the effect of extracorporeal shock wave therapy of gastrosoleus trigger points in patients with plantar fasciitis

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of plantar fasciitis
2. having at least one Gastrosoleus trigger point concomitantly.
3. having no response to conservative treatments for at least 3 months
4. willingness to participate

Exclusion Criteria:

1. Dysfunction of the knee or ankle
2. Neurologic abnormalities
3. Bleeding tendency (hereditary or acquired)
4. Nerve entrapment syndrome
5. A previous operation on the heel
6. Pregnancy
7. Evidences of Infection in lower limbs
8. A medical History of tumor
9. previous local corticosteroid injection within 12 weeks

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-08 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in pain severity after 3 weeks | Up to 4 weeks
  The pain score (100 mm Visual Analogue Score ) is evaluated before the first session and 4 weeks after the last session.

SECONDARY OUTCOMES:
Change from baseline in pain degree after 2 months. | Up to 2 months
  The pain score (100 mm Visual Analogue Score ) and the modified criteria of the Roles and Maudsley score are evaluated at baseline and then 2 months after therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Farnaz Dehghan, MD, Principal Investigator — Isfahan University of Medical Sciences
Locations (1):
- Department of Rehabilitation, Alzahra Hospital, Isfahan, Isfahan, Iran

REFERENCES:
- [Result] Wang CJ, Wang FS, Yang KD, Weng LH, Ko JY. Long-term results of extracorporeal shockwave treatment for plantar fasciitis. Am J Sports Med. 2006 Apr;34(4):592-6. doi: 10.1177/0363546505281811. PMID 16556754
- [Result] Cotchett MP, Landorf KB, Munteanu SE, Raspovic A. Effectiveness of trigger point dry needling for plantar heel pain: study protocol for a randomised controlled trial. J Foot Ankle Res. 2011 Jan 23;4:5. doi: 10.1186/1757-1146-4-5. PMID 21255460
- [Result] Gleitz M, Hornig K. [Trigger points - Diagnosis and treatment concepts with special reference to extracorporeal shockwaves]. Orthopade. 2012 Feb;41(2):113-25. doi: 10.1007/s00132-011-1860-0. German. PMID 22349369
- [Result] Ogden JA, Alvarez RG, Marlow M. Shockwave therapy for chronic proximal plantar fasciitis: a meta-analysis. Foot Ankle Int. 2002 Apr;23(4):301-8. doi: 10.1177/107110070202300402. PMID 11991474